CLINICAL TRIAL: NCT04035213
Title: Sleep, the Never-ending Quest of College Students: Effects of a Semester Long Sleep Course on Sleep Patterns and Daytime Functioning
Brief Title: Sleep, the Never-ending Quest of College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Simon Lau, Clinical Psychology Doctoral Candidate, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001775
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Sleep; Sleep Disturbance; Sleep Hygiene
MeSH Terms: conditions — Parasomnias; Sleep Hygiene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavior of Sleep Course (Experimental): A semester-long course focused on sleep improves college students' sleep patterns over one semester. The listed aims of this course are to: 1) provide students with a comprehensive understanding of sleep; 2) afford an overview of the multiple ways sleep impact health, performance and well-being; and 3) to assist students in discovering how their own sleep-wake patterns impact their day to day functioning.
  Interventions: Behavioral: Behavior of Sleep Course
- Control (No Intervention): Students from other upper level departmental courses with content that does not include a focus on or discussion of sleep

INTERVENTIONS:
Behavioral: Behavior of Sleep Course — The current study will evaluate whether a semester-long course focused on sleep improves college students' sleep patterns over one semester compared to students completing a similar-level course in the same department (Psychology) at the same university.
  Arms: Behavior of Sleep Course

SUMMARY:
The purpose of this study is to evaluate whether undergraduate students completing a course focused entirely on sleep at a major urban university evidence positive changes in their sleep patterns compared to students completing a similar-level course (without any discussion of sleep) in the same department (Psychology) at the same university (UH). Potential changes in sleep patterns across the semester will be examined as well as whether putative changes in sleep can be linked with academic and mental health outcomes.

DETAILED DESCRIPTION:
Aim 1) To evaluate whether a semester long course focused entirely on sleep produces improvements in college students' sleep patterns across the semester based on one-week sleep diaries.

H1: Compared to students enrolled in other courses who are not expected to show significant changes in sleep patterns, students enrolled in the sleep course will demonstrate increases in total sleep time, decreases in sleep onset latency, and decreases in nighttime awakenings. In line with Mayer's theoretical model, these sleep-based changes will evidence non-linear (i.e., quadractic) patterns across four time points during the semester.

Aim 2) To evaluate changes in sleep hygiene behaviors across the semester among students enrolled in a sleep course compared to students enrolled in other courses.

H2: Compared to students enrolled in other courses who are not expected to show significant changes in sleep hygiene behaviors, students enrolled in the sleep course will report a decreased frequency of naps, use of electronics within one hour of bed, and an increase in sleep regularity (e.g., reduction in the discrepancy between weekend and weekday wake times) across the four time points during the semester.

Aim 3) To evaluate how sleep patterns relate to daytime mood and energy levels across the semester among students enrolled in a sleep course and other courses.

H3: Greater total sleep time, shorter sleep onset latency, fewer nighttime awakenings, a less discrepancy between weekend and weekday wake times will predict higher energy levels and mood among both groups across the semester.

Aim 4) To evaluate how sleep patterns across the semester predict final course grades among students enrolled in a sleep course.

H4: Students enrolled in the sleep course who demonstrate increases in total sleep time, decreases in sleep onset latency, and decreases in nighttime awakenings across the semester will achieve higher final course grades than students who demonstrate minimal to no improvements in sleep.

ELIGIBILITY:
Inclusion Criteria:

* All undergraduate students at UH age 18 and older who are enrolled in the following upper-level courses and who provide consent to participate will be eligible to participate as control participants

Exclusion Criteria:

* Previous enrollment in PSYC 4397: The Behavior of Sleep course or a similar course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
National Sleep Foundation Sleep Diary | 7 days
  The National Sleep Foundation Sleep Diary is a self-report diary designed to help participants track their sleep, sleep habits, and other relevant sleep behaviors (e.g., caffeine use) over a seven-day period.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lau, M.A., Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No